CLINICAL TRIAL: NCT01130792
Title: Probiotics for Infectious Diarrhea in Children in South India
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Christian Medical College, Vellore, India (Other)
Collaborators: Indian Council of Medical Research (Other Government); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Tufts Medical Center (Other)
Responsible Party: Principal Investigator, Gagandeep Kang, Professor, Christian Medical College, Vellore, India
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: MCHPROBIO; R03HD057736 (NIH); CTRI/2010/091/000339 (Registry Identifier: Clinical Trials Registry of India)
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Infectious Gastroenteritis
Keywords: rotavirus; cryptosporidium; probiotics; intestinal function; immune response
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus GG (Experimental): LGG once daily for 4 weeks
  Interventions: Dietary Supplement: Lactobacillus GG
- Inulin (Placebo Comparator)
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Lactobacillus GG — 10 Billion Organisms Given Mixed In Milk As Food Supplement Once Daily For Four Weeks
  Arms: Lactobacillus GG
Dietary Supplement: Inulin — Identical appearing capsules containing a powder resembling the LGG to be given as for intervention
  Arms: Inulin

SUMMARY:
The overall goal of this study is to investigate whether the modulatory effects of probiotics, which are used as food supplements (Lactobacillus GG marketed as Culturelle or yoghurt) in the gastrointestinal tract promote restoration of intestinal function and enhance the specific immune response in children with cryptosporidial or rotaviral infections in South India. Rotavirus and Cryptosporidium spp. are the most important viral and parasitic causes of gastroenteritis in children in south India. Both infections can lead to severe dehydrating gastroenteritis in young children and have no specific treatment. Repeated episodes of diarrhea can result in long term deleterious effects on nutritional status, possibly due to intestinal damage. Most episodes of infectious gastroenteritis resolve without specific therapy, the mainstay of treatment being rehydration. However, oral rehydration remains under-utilized, in part due to the lack of effect on frequency of bowel movements and duration of illness. Due to the interest in simple, safe and effective measures to ameliorate the long-term effects of diarrheal illness, there is a growing appreciation for the potential of certain microorganisms to offer direct benefits to the health of a host. Probiotics are known to beneficially modulate several host functions, the most important of which are immune responses and intestinal barrier integrity. The investigators propose to build on the investigators previous collaborative efforts to conduct pilot studies to provide a mechanistic understanding of the effect of probiotic supplementation in children with rotaviral and cryptosporidial diarrhea.

Based on the established efficacy of LGG for the treatment of a variety of diarrheal diseases and the documented modulation of immune responses and strengthening of intestinal epithelial barrier function by probiotics, the investigators propose to conduct a Phase I/II double-blind randomized placebo controlled clinical trial to assess the preliminary efficacy and safety of LGG vs. placebo in the resolution of symptoms and restoration of intestinal function in children with either rotaviral or cryptosporidial diarrhea and no other detected enteric infection. Promising results in this Phase I/II study will provide preliminary data to power a future randomized trial on these critical outcomes following rotaviral or cryptosporidial infection.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children aged 6 months to 5 years
* Diagnosis of rotaviral or cryptosporidial gastroenteritis (Rotavirus or
* Cryptosporidium EIA positive and three or more watery stools within a 24-hour period)
* No other enteric pathogen isolated from the stool at the time of enrollment
* Able to take the contents of study capsules mixed into food or milk
* No need for antibiotics for current illness
* No use of LGG/other probiotics within 30 days (yogurt consumption is not an exclusion criterion)
* HIV negative
* No severe malnutrition (WAZ score < 3SD below the median)
* No evidence of active bowel leak, acute abdomen or colitis
* No history of allergy
* Parent/guardian willing to report on compliance and side effects during the study period
* Families willing to provide informed consent, participate in study and have study personnel visit their home.

Exclusion criteria

* Other enteric pathogens isolated from the stool at the time of enrollment
* Not willing or able to take the contents of study capsules mixed into food or milk
* Need for antibiotics for current illness
* HIV positive
* Severe malnutrition (WAZ score < 3SD below the median)
* Presence of active bowel leak, acute abdomen or colitis
* History of allergy
* Parent/guardian not willing to report on compliance and side effects during the study period
* Families not willing to provide informed consent, participate in study or have study personnel visit their home.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
IgG To Rotavirus VP6 Or Cryptosporidial Gp15 | 4 weeks

SECONDARY OUTCOMES:
lactulose:mannitol test | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gagandeep Kang, MD, PhD, Principal Investigator — Christian Medical College, Vellore, India; Honorine D Ward, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Christian Medical College, Vellore, Tamil Nadu, India

REFERENCES:
- [Result] Sindhu KN, Sowmyanarayanan TV, Paul A, Babji S, Ajjampur SS, Priyadarshini S, Sarkar R, Balasubramanian KA, Wanke CA, Ward HD, Kang G. Immune response and intestinal permeability in children with acute gastroenteritis treated with Lactobacillus rhamnosus GG: a randomized, double-blind, placebo-controlled trial. Clin Infect Dis. 2014 Apr;58(8):1107-15. doi: 10.1093/cid/ciu065. Epub 2014 Feb 5. PMID 24501384